CLINICAL TRIAL: NCT03638557
Title: The Effect of School Lunch Program (SLP) Towards Nutrition Knowledge, Attitude, Practices and Nutrition Status of Adolescents in Islamic Boarding School
Brief Title: School Lunch Program (SLP) Towards Nutrition Knowledge, Attitude, Practices and Nutrition Status of Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Pertanian Bogor (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Reisi Nurdiani, SP, MSi, Secretary of Department of Community Nutrition, Institut Pertanian Bogor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SLP05/2018
Record Dates: First submitted 2018-08-06; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Anemia; Stunting; Underweight
MeSH Terms: conditions — Anemia; Growth Disorders; Thinness

STUDY DESIGN:
Intervention Model Description: pre-post quasi experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention package consists of the following;
  1. Balanced Nutrition and Clean and Healthy Lifestyle Behavior Education for the boarding school students (once a week with the duration of 30-60 minutes. 3 weeks are delivered by trained teachers, and 1 week by research team.
  2. Nutritious lunch, for 7 days a week. With the total of 220 days. The lunch menu is designed to meet 30% of the students RDA, which consists of 635-777 Kcal and 18-22 grams of protein
  Interventions: Other: Nutritious Lunch

INTERVENTIONS:
Other: Nutritious Lunch — The intervention package consists of the following;
  1. Balanced Nutrition and Clean and Healthy Lifestyle Behavior Education for the boarding school students (once a week with the duration of 30-60 minutes. 3 weeks are delivered by trained teachers, and 1 week by research team.
  2. Nutritious lunch, for 7 days a week. With the total of 220 days. The lunch menu is designed to meet 30% of the students RDA, which consists of 635-777 Kcal and 18-22 grams of protein

SUMMARY:
The main objective of this study is to assess the impact of the school lunch program and nutrition education towards the change in knowledge, attitude, and behavior on balanced nutrition and clean and healthy lifestyle behavior (CHLB) of adolescents living in an Islamic Boarding School. The secondary objective is to assess the program impact on energy and nutrient intake, nutrition status, hemoglobin concentration, physical fitness and concentrating ability of students.

A pre-post quasi experimental design is applied to assess the impact. The intervention includes: 1) provision of nutritious lunch, meeting the nutrient requirements of adolescents for one meal, for 7 days a week, with the total duration of 220 days, 2) provision of nutrition education once a week (3 times delivered by teachers, 1 time delivered by research team) and nutrition education media, 3) capacity building of teachers and food handlers. The duration of the intervention is 1 academic year or 8 active months after the reduction of holidays and examination months.

DETAILED DESCRIPTION:
This research will be conducted using pre-post quasi experimental design. Subjects consist of only intervention group, who are measured before and after the intervention or program period. The SLP program (intervention) in Darussalam Islamic Boarding School consists of:

1. Balanced Nutrition Education and CHLB for the boarding school students and teachers
2. Provision of lunch
3. Food processing training, food sanitation hygiene and food safety for food handlers.

The location of this activity is determined purposively at the Islamic boarding school, in the neighborhood of the IPB (Institut Pertanian Bogor) campus with the following basic criteria for the school:

1. Has apparent nutritional problems among the students
2. It has a kitchen and dining area for its students in need of improvement
3. Has a strong commitment to cooperate in running the program. This activity will be held at the Darussalam Islamic Boarding School located in Laladon Bogor area. There are 450 students consisting of both male and female students. This Islamic boarding school has a kitchen that is used to process and cook food for the students. The eating area is divided into two areas, in the form of a shared dining room for the male students and a terrace for the female students. The Islamic boarding school also has a garden area that is used for gardening activities for the students but it has not been managed in a sustainable manner.

The overall project period is 18 months (2017/09-2019/03), which includes design, baseline, midline and endline data collection (3 times), implementation and reporting activities. The implementation of the school lunch program will be for 1 academic year (8 active months after the reduction of holidays and examination months), starting immediately after Institutional Review Board (IRB) approval of both Bogor University and Ajinomoto co. inc.until the end of March 2019. Lunch will be served 7 days per week with the total of 220 days The provision of lunch is designed to meet 30% of the daily nutritional requirements of students and contains 635-776 Kcal of energy with 18-22 grams of protein. The lunch menu is served in the form of a full menu consisting of staple food, animal products, plant products, vegetables and fruit by utilizing local food. The menu cycle used is a set menu cycle of 10+1 day cycle Hemoglobin level and dietary intake data was collected for sub sample of students, meeting the sample size calculation, which was 150 subjects. Data will be collected at baseline (before the intervention), midline, and endline.

ELIGIBILITY:
Inclusion Criteria:

* have resided in the boarding school at least one year
* are anemic or underweight or stunted

Exclusion Criteria:

* severely anemic with Hb concentration < 7 g/dl
* BMI for age z-score <-3

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin concentration using Hemocue | February-November (9 months)
  Hemoglobin concentration of subjects measured using Hemocue

SECONDARY OUTCOMES:
Body Mass Index (BMI) for age z-score | February-November (9 months)
  Indicator of nutrition status of adolescents, measured by the assessment of weight and height of the subject. BMI for age z-score was calculated using World Health Organization (WHO) Anthro Plus Software
Nutrition and health knowledge using validated-structured questionnaire | February-November (9 months)
  Knowledge on nutrition and clean and healthy lifestyle behavior
Nutrition and health practices using validated-structured questionnaire | February-November (9 months)
  Practices related to nutrition and clean and healthy lifestyle behavior
Nutrition and health attitude using validated-structured questionnaire | February-November (9 months)
  Attitude on nutrition and clean and healthy lifestyle behavior (values of subjects), measured by questionnaire asking whether they agree or disagree to statements on nutrition and health
Nutrient intake using Semi Quantitative Food Frequency Questionnaire | February-November (9 months)
  Energy, protein, carbohydrate, fat, iron, zinc, and vitamin c intake. Assessed using 24 hour recall
Food pattern using validated-structured questionnaire | February-November (9 months)
  Consumption of protein sources, vegetables, fruits, dairy products and beverages. Assessed using Food Frequency Questionnaire
Physical Fitness based on the Indonesian Physical Fitness Test | February-November (9 months)
  A series of test using the Indonesian Physical Fitness Test, consisting of push up, sit up, high jump, sprint, and running 1000 m
Concentration/ short term memory using memory cards based on Kustiyani 2005 | February-November (9 months)
  Assessed using a set of cards to memorize with reduced duration of time

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rimbawan, Principal Investigator — Department of Community Nutrition, Faculty of Human Ecology, Bogor Agricultural University
Locations (1):
- Darussalam Islamic Boarding School, Bogor, West Java, Indonesia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT03638557/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT03638557/ICF_001.pdf